CLINICAL TRIAL: NCT06089824
Title: Drug Utilisation and Safety Study of Mysimba in Europe and Contrave in the United States
Brief Title: Drug Utilisation of Mysimba/Contrave
Acronym: DUS
Status: Completed | Type: Observational
Sponsor: Currax Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: NB-451
Record Dates: First submitted 2023-10-12; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will assess a retrospective cohort of users of Mysimba/Contrave with up to 548 days (~18 months) after initiation with treatment with Mysimba/Contrave. This study will describe Mysimba/Contrave utilisation and incidence of AESIs for users compliant and non-compliant with the SmPC.

ELIGIBILITY:
Inclusion Criteria:

* At least one prescription of Mysimba/Contrave in his/her medical records any time during the study period (US) OR at least one dispensing of Mysimba/Contrave in his/her registry any time during the study period (Nordic);
* At least 365 days of computerized records prior to first Mysimba/Contrave prescription or dispensing date; and3Patient is active (i.e., alive and registered/accruing data) at the time of the first Mysimba/Contrave prescription or dispensing date.

Exclusion Criteria:

- All patients meeting inclusion criteria will be included in the study; no exclusion criteria will be applied.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Users of Mysimba/Contrave with at least 365 days of computerized records prior to first use in Denmark Finland, Norway and Sweden, and other countries (if meeting the threshold for patients and agreed upon between EMA and MAH) with sufficient uptake of Mysimba/Contrave in the respective national health systems. Additionally, U.S. data will be included.
Sampling Method: Non-Probability Sample
Enrollment: 43324 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2022-10 (Actual); Study Completion 2022-10 (Actual)

PRIMARY OUTCOMES:
Demographic characteristics of patients initiating use of Mysimba/Contrave (Age) | All available follow-up data up to 548 days after the index date will be included for each patient or end of study period
  Patient demographics (years of age on index date)
Demographic characteristics of patients initiating use of Mysimba/Contrave (Sex) | All available follow-up data up to 548 days after the index date will be included for each patient or end of study period
  Patient demographics (sex [male/female] on index date)
Demographic characteristics of patients initiating use of Mysimba/Contrave (Race) | All available follow-up data up to 548 days after the index date will be included for each patient or end of study period
  Clinically recorded race (i.e., White, Black or African American, Asian, or other/unknown) and ethnicity (i.e., Hispanic or Latino, Non-Hispanic or Latino, or unknown)
Demographic characteristics of patients initiating use of Mysimba/Contrave (Smoking Status) | All available follow-up data up to 548 days after the index date will be included for each patient or end of study period
  Smoking status (i.e., current or ever)
Demographic characteristics of patients initiating use of Mysimba/Contrave (Comorbidities) | All available follow-up data up to 548 days after the index date will be included for each patient or end of study period
  Existing comorbidities:
  * Metabolic comorbidities (i.e., diabetes or dyslipidemia);
  * Hypertension;
  * Seizure disorder;
  * Hepatic impairment;
  * Central nervous system tumor
Demographic characteristics of patients initiating use of Mysimba/Contrave (Substance Abuse/Dependencies) | All available follow-up data up to 548 days after the index date will be included for each patient or end of study period
  History of substance abuse/dependencies; including acute opioid withdrawal
Demographic characteristics of patients initiating use of Mysimba/Contrave (Medical Conditions) | All available follow-up data up to 548 days after the index date will be included for each patient or end of study period
  History of the following medical conditions:
  * Seizures;
  * Bipolar disorder;
  * Major depressive disorder (MDD);
  * Anorexia nervosa;
  * Bulimia;
  * Prior use of naltrexone, bupropion, opioid, or MAOI
Demographic characteristics of patients initiating use of Mysimba/Contrave (Pregnancy) | All available follow-up data up to 548 days after the index date will be included for each patient or end of study period
  Pregnancy status.
Demographic characteristics of patients initiating use of Mysimba/Contrave (Breastfeeding) | All available follow-up data up to 548 days after the index date will be included for each patient or end of study period
  Breastfeeding status.
Patterns of Mysimba/Contrave initiation (Rx) | All available follow-up data up to 548 days after the index date will be included for each patient or end of study period
  Mysimba/Contrave initiation includes number of prescriptions
Patterns of Mysimba/Contrave initiation (Episodes) | All available follow-up data up to 548 days after the index date will be included for each patient or end of study period
  Mysimba/Contrave initiation includes number of treatment episodes
Patterns of Mysimba/Contrave initiation (Duration) | All available follow-up data up to 548 days after the index date will be included for each patient or end of study period
  Mysimba/Contrave initiation includes duration between prescriptions
Baseline characteristics of patients initiating use of Mysimba/Contrave (Height) | All available follow-up data up to 548 days after the index date will be included for each patient or end of study period
  Height (meters) (most recent value on or before the index date)
Baseline characteristics of patients initiating use of Mysimba/Contrave (Weight) | All available follow-up data up to 548 days after the index date will be included for each patient or end of study period
  Weight (kg) (most recent value on or before the index date)
Baseline characteristics of patients initiating use of Mysimba/Contrave (BMI) | All available follow-up data up to 548 days after the index date will be included for each patient or end of study period
  BMI (kg/m2) (most recent value on or before the index date) (obtained directly from data sources; BMI may be calculated if height and weight available)
Patterns of Mysimba/Contrave use (Compliance) | All available follow-up data up to 548 days after the index date will be included for each patient or end of study period
  Mysimba/Contrave use includes the number and percentage of patients compliant with the SmPC.
Patterns of Mysimba/Contrave use (Non-compliance) | All available follow-up data up to 548 days after the index date will be included for each patient or end of study period
  Mysimba/Contrave use includes the number and percentage of patients non-compliant with the SmPC.

CONTACTS AND LOCATIONS:
Locations (1):
- Currax Pharmaceuticals, Nashville, Tennessee, United States